CLINICAL TRIAL: NCT00001252
Title: A Rigid Body Database on Human Movement
Brief Title: Human Movement Database
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 900168; 90-CC-0168
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Movement Disorder
Keywords: Biomechanics; Kinesiology; Walking; Natural History
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteer: Normal/healthy volunteers
- Impaired volunteer: volunteers with impairments of the neuromusculoskeletal system.

SUMMARY:
This study will collect information on the different ways people control limb and body movements. This information will be used to develop a database on normal movements and adaptive movements of people who have diseases that affect the way they move. The database will serve as a tool to improve diagnosis and treatment of patients with movement-related problems.

Volunteers from one month old to old age who have normal movement patterns or who have developed different ways to perform movement tasks may be eligible for this study. A physician or physical therapist will screen candidates to determine their strength, flexibility and range of motion of joints.

Participants will be asked to perform movements such as walking, walking up or down stairs, standing quietly or reaching for an object or using treadmill. For the test, the arms and legs are wrapped with a soft, rubber-like material to which small plastic reflective balls are attached. A piece of firm material called a shell may be attached to the rubber sleeves or other areas of the body. Then the volunteer performs the specified task several times while special cameras record the movement. These cameras will record the positions of the reflective balls during movement and may show the person s face or body. Electrical activity in the muscles also may be measured, using small metal electrodes attached to the surface of the skin with an adhesive bandage.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

The purpose of this study is to develop a database of normative and adaptive control strategies for human motion. Volunteers will serve as subjects after they complete a neuromusculoskeletal screening exam. Subjects will be asked to perform one or more tasks related to the execution of activities of daily living such as: walking on the ground, walking on a treadmill, quiet and perturbed standing, stair ascent and descent, turning and jumping, and isolated upper and lower extremity limb movements or trunk movements. The subjects movement patterns will be recorded using a three-dimensional motion tracking system. Motion data will be analyzed using a rigid body six degree-of-freedom approach when applicable. Temporal/spatial, kinematic, kinetic, and surface electromyographic variables will be collected and calculated. When only temporal-spatial parameters are of interest, an instrumented portable walkway system may be used.

OBJECTIVES:

Primary objectives:

To develop a database of normative and adapted movement strategies for human movement. The variables calculated from the established database will be presented as mean time histories to serve as standards by which individual patient and group motion data may be compared.

ENDPOINTS:

Primary Endpoint:

The primary endpoint here is to accumulate a large database of participants with and without different neuromuscular disorders that includes multiple measures of physical function and performance, so we can begin to investigate the mechanisms underlying various disorders on either a group or individual basis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals with neuromuscular disorders and Healthy Volunteers in order to be eligible to participate in this study, must meet all of the following criteria:

* Children; One month old to 17 years of age

  --In the case of infants and very young children, they need to be able to imitate or perform an action on cue (e.g., reach out for a toy that is presented or take steps if placed on a treadmill) based on the parent report if the subject is a child and physician observation during history and physical examination.
* Adults; 18 years 99 years
* In good general health as evidenced by medical history or diagnosed with impairment of neuromusculoskeletal system
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Provision of signed and dated informed consent form
* For those participants older than 5 years of age who have an abnormal gait pattern when walking as a result of a central nervous system injury, Dr. Alter will ask them or their guardian about their seizure history

EXCLUSION CRITERIA:

Individuals with neuromuscular disorders and Healthy Volunteers, who meets any of the following criteria will be excluded from participation in this study:

* Individuals with pacemakers
* Pregnancy
* Adults unable to provide informed consent

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal/healthy volunteers and volunteers with impairments of the neuromusculoskeletal system. Subjects will be evenly distributed between males and females
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 1995-03-13 (Actual)

PRIMARY OUTCOMES:
Gait Kinematics | end of testing
  Strength and spasticity testing both include torque or force measurements as the primary outcomes. Balance testing typically yields the amount, velocity and direction of sway in response to different conditions or perturbations.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine E Alter, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on IPD sharing.

REFERENCES:
- [Background] Murray MP. Gait as a total pattern of movement. Am J Phys Med. 1967 Feb;46(1):290-333. No abstract available. PMID 5336886
- [Background] Benvenuti F, Stanhope SJ, Thomas SL, Panzer VP, Hallett M. Flexibility of anticipatory postural adjustments revealed by self-paced and reaction-time arm movements. Brain Res. 1997 Jun 27;761(1):59-70. doi: 10.1016/s0006-8993(97)00260-6. PMID 9247066
- [Background] Hallett M, Lebiedowska MK, Thomas SL, Stanhope SJ, Denckla MB, Rumsey J. Locomotion of autistic adults. Arch Neurol. 1993 Dec;50(12):1304-8. doi: 10.1001/archneur.1993.00540120019007. PMID 8257307
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1990-CC-0168.html